CLINICAL TRIAL: NCT06426290
Title: Prediction of Response to Bariatric Surgery Treatment in Patients Suffering From Severe Obesity, Based on the Scales of the MMPI-2-RF Questionnaire Carried Out Preoperatively
Brief Title: Prediction of Response to Bariatric Surgery in Patients With Severe Obesity
Acronym: PREDI-CHIRBA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Moulins Yzeure (Other)
Responsible Party: Sponsor
Other Study IDs: CHMY-2021-06
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: post-surgery psychological evaluation — Following questionnaires will be done :
  Patient Health Questionnaire (PHQ-9) Generalized Anxiety Disorder (GAD-7) Three Factor Eating Questionnaire (TFEQ-R21) Quality of life for obesity and dietetic questionnaire (EQVOD) Body Esteem Scale (BES) Figure Rating Scale (auto-questionnaire)

SUMMARY:
This is an retrospective and prospective (ambispective) study with data collection from volunteer patients who passed an MMPI-2-RF (Minnesota Multiphasic Personality Inventory-2-Restructured form) questionnaire in the preoperative phase of a bariatric surgery project.

The evolution of their BMI will be correlated to psychological dimensions collected in patient questionnaires, before and after bariatric surgery.

The presence of possible risk factors such as depression, anxiety, eating disorders, quality of life, satisfaction and the perception of body, could make it possible to establish adapted therapies before surgery, in order to attenuate or eliminate the presence of these factors, and improve BMI evolution and bariatric surgery success.

DETAILED DESCRIPTION:
A first phase of data collection will concern data from the MMPI-2-RF questionnaire as well as clinical data, collected during preoperative consultations.

For the second phase, post-operative data will be collected, during a routine follow-up consultation in the nutrition Department, where specific psychological questionnaires are taken by patients.

ELIGIBILITY:
Inclusion Criteria:

* Having been treated in the Nutrition department for severe obesity and considered for bariatric surgery because having met the criteria validating bariatric surgery:
* Having passed the MMPI-2-RF questionnaire between January 1, 2014 and December 31, 2023 in the preoperative phase, as part of psychological follow-up
* Having benefited from bariatric surgery or patients who have abandoned the surgery plan for a reason other than a medical contraindication.
* Informed of the study, having agreed to participate and not having opposed the use of their data

Exclusion Criteria:

* Subjects who generated an invalid MMPI-2-RF questionnaire, according to the test validity criteria (verified by the principal investigator)
* Subjects who expressly objected to the use of their data for this study
* Subjects who have not undergone bariatric surgery due to a medical contraindication.
* Patient unable to understand the study or complete the post-operative phase visit
* Persons under guardianship or curators or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe obesity : BMI > 40 kg/m2 or > 35 kg/m2 associated with at least one comorbidity likely to be improved after surgery.
  * Failure of well-conducted medical, nutritional, dietetic and psychotherapeutic monitoring for 6-12 months
  * Lack of sufficient weight loss or failure to maintain weight loss
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine the predictive value of depressive symptomatology dimension on the evolution of BMI. | At inclusion psychological consultation
  Depressive dimension assessed by the preoperative MMPI-2-RF questionnaire and compared to the same dimension from post-surgery psychological questionnaires.

SECONDARY OUTCOMES:
Determine the predictive value of anxiety symptomatology dimension on the evolution of BMI | At inclusion psychological consultation
  Anxiety dimension assessed by the preoperative MMPI-2-RF questionnaire and compared to the same dimension from post-surgery psychological questionnaires.
Determine the predictive value of eating behavior dimension on the evolution of BMI | At inclusion psychological consultation
  Eating behaviour dimension assessed by the preoperative MMPI-2-RF questionnaire and compared to the same dimension from post-surgery psychological questionnaires.
Determine the predictive value of quality of life dimension on the evolution of BMI | At inclusion psychological consultation
  Quality of life dimension assessed by the preoperative MMPI-2-RF questionnaire and compared to the same dimension from post-surgery psychological questionnaires.
Determine the predictive value of satisfaction and body perception dimensions on the evolution of BMI | At inclusion psychological consultation
  satisfaction and body perception dimensions assessed by the preoperative MMPI-2-RF questionnaire and compared to the same dimension from post-surgery psychological questionnaires.
Determine typical profiles of patients who have finally denied surgery apart from medical contraindications | At inclusion psychological consultation
  Using the MMPI-2-RF preoperative questionnaire
Identify the risk factors for abandonment or difficulties after the intervention, in order to establish appropriate preoperative treatments before surgery | At inclusion psychological consultation
  Using the MMPI-2-RF preoperative questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Virginie ALLASSEUR, psychologist, Principal Investigator — Centre Hospitalier de Moulins Yzeure
Locations (1):
- Centre hospitalier Moulins-Yzeure, Moulins, France